CLINICAL TRIAL: NCT05724966
Title: Anti-neoplastic Treatment, Based on PRO Data Reported Through a MHealth App Solution in Multiple Myeloma - a Mixed Method Study
Brief Title: Anti-neoplastic Treatment, Based on PRO Data Reported Through a MHealth App Solution in Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Thomas Lund (Other)
Responsible Party: Sponsor-Investigator, Thomas Lund, MD, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: Fit for treatment
Record Dates: First submitted 2023-01-09; First posted 2023-02-13 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Registration of side effects: patients are to registrer side effects prior to treatment with Bortezomib through an app.
  Interventions: Device: mHealth app

INTERVENTIONS:
Device: mHealth app — We wish to examine the perspectives of patients with multiple myeloma and healthcare professionals of this new method for reporting side effects, and to assess organizational aspects. Usual procedure to assess side effect prior to cancer treatment with Bortezomib is a telephone call the day before.

SUMMARY:
Pirmary endpoint: to examine the feasibility of using an mHealth app for reporting of side effects instead of a telephone call from the hospital staff together with examining the perspectives of patients with multiple myeloma and healthcare professionals of this new method for reporting side effects, and to assess organizational aspects. Usual procedure to assess side effect prior to cancer treatment with Bortezomib is a telephone call the day before. With this innovative method investigator aimed to give the patient more independence in their daily life and in that way improve their quality of life.

DETAILED DESCRIPTION:
It is a prospective, clinical, parallel mixed-method design with a quantitative core and a qulitative supplementary component. There will be used a Mhealth app called "My Hospital".

Quantitative data will be acquired from time registrations performed by patients and nurses and will be descriptively analyzed applying a micro-costing approach, using cost data per individual. Qualitative data will be obtained from individual, semi-structured interviews with patients and one focus group interview with healthcare professionals and will be analyzed applying a hermeneutic approach.

Eligible for inclusion were patients with MM scheduled for Bortezomib. Moreover, patients should have access to a smartphone, be able to self-report side effects of Bortezomib using a smartphone app, and be willing to participate in a semi-structured interview.

ELIGIBILITY:
Inclusion Criteria:

* patients with MM scheduled for Bortezomib
* patients should have access to a smartphone
* patients should be able to self-report side effects of Bortezomib using a smartphone app, and be willing to participate in a semi-structured interview.

Exclusion Criteria:

* patients had to talk and read danish

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Myeloma planned treatment with Bortezomib.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Time registrations of side effects using an app | 18 months
  PRO data (time registrations of side effects using an app)
patient registration of side effects using an app | 18 months
  PRO data

SECONDARY OUTCOMES:
Qualitative perspectives interview | 16 months
  Through semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Jannie Kirkegaard, RN, Principal Investigator — Odense Universitetshospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No